CLINICAL TRIAL: NCT01598389
Title: Eating Behaviors Among Weight-Discordant Siblings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tanja Kral, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: K01DK078601 (NIH)
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low energy-dense preload (Experimental)
  Interventions: Other: Feeding study
- High energy-dense preload (Experimental)
  Interventions: Other: Feeding study
- No preload (Experimental)
  Interventions: Other: Feeding study

INTERVENTIONS:
Other: Feeding study — In a crossover design, siblings were served dinner once a week for 3 weeks. Across conditions, siblings were served the same dinner, but, 25 minutes before dinner, they either consumed in full or did not consume one of two preloads that varied in energy density. On the day when no preload was consumed, eating in the absence of hunger was assessed after dinner and defined as the number of calories consumed from snacks. Habitual dietary intake was assessed using 24-hour dietary recalls.

SUMMARY:
The purpose of this study was to compare weight-discordant siblings in eating in the absence of hunger, caloric compensation, and the quality of their habitual diet. The investigator hypothesized that, within families and controlling for age differences, overweight and obese siblings would show greater eating in the absence of hunger, poorer caloric compensation, and poorer diet quality (e.g., increased percent of energy from fat and caloric beverages) compared to normal-weight siblings.

DETAILED DESCRIPTION:
The study used a discordant sibling design to compare putative obesity-promoting eating traits among siblings, 5-12 years, who were raised in the same household, but were discordant for weight status (normal-weight: BMI-for-age between 5 and less than the 85th percentile; overweight/obese: BMI-for-age greater or equal to the 85th percentile). Forty-seven pairs of same-sex siblings (boys and girls) were recruited from the greater Philadelphia area to participate in a 4-week study during which their eating behaviors and body composition were assessed. The study tested the hypotheses that overweight/obese, compared to normal-weight, siblings exhibit 1) a weaker ability to compensate for calories, 2) a greater susceptibility towards eating in the absence of hunger, and 3) habitual dietary intakes that favor increased dietary energy density (kcal/g) and increased %energy derived from fat and caloric beverages. The use of a behavioral genetics design to study eating phenotypes among siblings is a unique approach to elucidate shared and non-shared environmental influences that can contribute to variations in weight status during childhood.

ELIGIBILITY:
Inclusion Criteria:

* same-sex;
* weight discordant (normal-weight vs. overweight/obese);
* meet age criteria;
* like most foods that were served in the study.

Exclusion Criteria:

* serious medical conditions or medication use known to affect appetite, food intake and body weight;
* developmental or psychiatric conditions;
* food allergies or nutrient intolerances (including lactose intolerance).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Energy intake | Up to 4 weeks
  %COMPX, EAH, dietary intake variables

SECONDARY OUTCOMES:
Body composition | Single assessment at Week 4
  Weight status (BMI-for-age percentile), BMI z-score, total body fat (%), waist circumference (cm), skinfold thickness (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja V.E. Kral, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kral TV, Allison DB, Birch LL, Stallings VA, Moore RH, Faith MS. Caloric compensation and eating in the absence of hunger in 5- to 12-y-old weight-discordant siblings. Am J Clin Nutr. 2012 Sep;96(3):574-83. doi: 10.3945/ajcn.112.037952. Epub 2012 Aug 1. PMID 22854400
- See also: National Institute of Diabetes and Digestive and Kidney Diseases — http://www2.niddk.nih.gov/